CLINICAL TRIAL: NCT03550976
Title: The Effect of Early Nutrition Intervention on the Incidence of High-risk Patients With Gestational Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Liuyanping, Clinical Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: hs-1551
Record Dates: First submitted 2018-05-29; First posted 2018-06-11 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High risk intervention group (Experimental)
  Interventions: Behavioral: The low-GI diet and muscle training
- High risk control group (No Intervention): Dietary evaluation and body composition analysis at 12 and 28 weeks of pregnancy. Receive routine obstetric examinations and routine health education which includes proper diet and exercise advice.Collect birth outcomes.
- Low risk control group (No Intervention): Dietary evaluation and body composition analysis at 12 and 28 weeks of pregnancy. Receive routine obstetric examinations and routine health education which includes proper diet and exercise advice.Collect birth outcomes.

INTERVENTIONS:
Behavioral: The low-GI diet and muscle training — During the 12-28 weeks of pregnancy, the pregnant women received low-GI diet and exercise intervention.Every two weeks, the pregnant women were followed up to assess the dietary situation and analyze the body composition results.Collect birth outcomes
  Arms: High risk intervention group

SUMMARY:
The incidence of gestational diabetes increased.The multidisciplinary management of GDM during pregnancy is helpful to improve the pregnancy outcome, but it will occupy huge medical resources.Early prediction, diet and exercise interventions can reduce the incidence of gestational diabetes, but there is no reliable way to predict and intervene early.This study is a randomized controlled trials, and aims to use comprehensive prediction method (genetic screening, body composition, clinical risk factors screening) screening the subjects with high GDM risk in early pregnancy, conducting diet and exercise intervention in second trimester and observing the effect on the incidence of GDM and perinatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* early pregnant women (< 12 weeks)
* fasting blood glucose < / = 5.6 mmol/L and glycosylated hemoglobin < / = 5.6%
* prepregnancy overweight (BMI > 23.9) or body fat content more than 30% (based on body composition analysis)
* no history of major diseases or long-term drug treatment
* no obvious physical disabilities, the ability of physical activity is normal
* dietary behavior and mental is normal
* resident in Beijing, early and middle stage pregnancy can be in Beijing area to receive regular obstetric examinations
* signed informed consent
* the following at least one

  * first-degree relatives family history of diabetes
  * history of abnormal lipid metabolism or abnormal lipid metabolism
  * history of polycystic ovary syndrome
  * history of large for gestational age infant or macrosomia deliver

Exclusion Criteria:

* history of gestational diabetes mellitus
* clinical glucose metabolism abnormalities
* once taking diabetes drugs or insulin injections
* a variety of food allergies or food choices serious limitations
* exercise during pregnancy contraindication

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-09-10 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of gestational diabetes | 12-28 weeks of pregnancy
  The incidence of GDM was compared between the low-GI diet and the muscle training group, the high-risk control group and the low-risk control group.